CLINICAL TRIAL: NCT04883086
Title: Holistic Approach to Investigate Protective and Risk Factors for Dental Caries in Patients With or Without Diabetes Type 2
Brief Title: Are Diabetics Type 2 More Prone to Dental Caries?
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: The Novo Nordisk UK Research Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 261531
Record Dates: First submitted 2020-11-23; First posted 2021-05-12 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus, Type 2; Dental Caries
Keywords: dental caries; oral health; diabetes; dental caries risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dental Caries; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — 1. Unstimulated and stimulated whole saliva collected by spitting technique.
  2. Blood sample carried out by a registered nurse.
  3. Supragingival plaque collection.
  4. Extracted teeth for laboratory resear
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic group ( Case): Total of 91 participants diagnosed with diabetes type 2
- Non diabetic group (control): Total of 91 participants healthy and not diagnosed with diabetes Mellitus

SUMMARY:
Background: Diabetes mellitus (DM) is well known for long-term complications to general and oral health. Periodontal disease has a bidirectional association with the development of type 2 diabetes (T2DM) (Mealey, 2006; Taylor, 2001; Demmer et el.,2008). However, current literature conflicts with regards to dental caries incidence in patients with T2DM (Sampaio, Mello and Alves, 2011).

Objective: To investigate potential protective and risk factors for dental caries among T2DM with vitamin D and HbA1c using clinical, salivary and microbial analyses.

Methods: This project is a case-control clinical study. The study will be conducted at Royal London Dental Hospital, Institute of Dentistry, Bart's Health NHS Trust, London, UK. This study will aim to recruit 182 participants in total with diabetes (type 2), aged ≥18 male or female and participants will be cross-matched with non-diabetes according to age and gender.

Each participant will undergo a baseline screening for around 60 minutes where all the following assessments will be carried out; Caries risk assessment (CAMBRA), Plaque index, International Caries Detection and Assessment System (ICDAS) and Laser fluorescence evaluator (SOPRLIFE®, Acteon, France) and Oral behavioural and sociodemographic background will be collected.

Prior to the clinical study, there will be a laboratory based study using extracted teeth. The aim of this ex-vivo study is to assess the autofluorescence variation in dental carious lesions and compare this with International Caries Detection and Assessment System (ICDAS).

DETAILED DESCRIPTION:
Research purpose:

The research question is individuals with Diabetes Mellitus type 2 (T2DM) is more prone to dental caries?

Several literature reviews point the lack of solid evidence clear association of the DM and dental caries (Ship, J.A., 2003; Taylor et al., 2004; Lamster, I.B., 2014; Garton et al., 2012; Leite et al., 2013).Also, a controversial result available of the epidemiology of dental caries among individuals with T2DM (Sampaio, Mello and Alves, 2011), besides limited knowledge about the biological explanation as seen with periodontal disease (Verhulst et al., 2019).Moreover, no study had a comprehensive evaluating of all potential caries risk factors. Thus this study developed a preliminary conceptual model in which 48 potential risk factors were identified and categorised into four domains: biological/intra-oral factors, medical factors, oral health behaviour, and sociodemographic factors.

All these potential factors will be evaluated and analysed through different appoaches; clinical, salivary, microbial analyses and patient questionnaire.

Recruitment process:

All participants (n=182) who meet the selection criteria and agree to participate will be invited to complete written informed consent by the PI.

Invitation letters will be sent by the DARE database holders to Diabetes patients who are on this database. Diabetes patients from Royal London Dental Hospital including outreach centres (Barkantine, Southend and Guttman), General Endocrinology and Metabolic Medicine, Diabetic clinics (including Mile End hospital) will also be invited using another invitation letter.

Regarding the control group, adult patients attending Dental Institute including outreach centres (Barkantine, Southend and Guttman), staff within Queen Mary University of London and Barts Health Trust and volunteers who agree to participate will be recruited.

All these participants will be approached and asked by the PI/CI whether they would be interested in taking part in this research. Participants who meet the inclusion criteria, will receive a written Patient Information Sheet (PIS) describing the study in details (Appendix 3). Subsequently, they will be asked by the Principal Investigator (AA) to complete and sign written informed consent (Appendix 4), if they wish to take part in this study. This phase will take around 15 minutes.

Those who consent to take part will be given an appointment to attend the dental clinic for assessments at the Institute of Dentistry.

Participants may enter the trial if the following apply:

* Participants who are male or female ≥ 18 years of age.
* For the test group, they have been diagnosed with type 2 Diabetes
* For the control group, participants who are not diagnosed with type 2 Diabetes
* Particiapants having minimum one natural tooth
* They are capable of giving informed consent
* They have the ability to understand and speak English
* They are able and willing to comply with all trial requirements
* They are not participating in another dental trial
* They are not diagnosed for cognitive defect due to mental illness, depression, Alzheimer's disease, or dementia.
* No antibiotic, no steroidal and/or non-steroidal anti-inflammatory medication used during the last 3 weeks
* Participants who are not pregnant and also not breastfeeding
* Participations who are not in another dental study testing different dental products during the previous three months and during the study period
* Participants who are not currently taking Vitamin D supplements

Exclusion criteria

* Participants who are edentulous
* Cognitive defect due to mental illness, depression, Alzheimer's disease, or dementia.
* The presence of any hard or soft tissue tumours in the oral cavity
* Patients undergoing chemo and/or radiation therapy
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Any condition, which in the opinion of the investigator, would preclude participation by the subject (such as cross-infection control risk)
* Participants who are prescribed long-term systematic antibiotics
* Participants who are pregnant and breastfeeding
* Participations who are in another dental study testing different dental products during the previous three months and during the study period
* Participants who had additional fluoride treatment in the past 6/3 months
* Participants who are prescribed to use high fluoridated toothpaste
* Participants who are currently taking Vitamin D supplements

Consent:

The potentially capable participant will be asked to confirm that they:

1. Read and understand the information sheet for the study.
2. Had the opportunity to consider the information, ask questions and have had these answered satisfactorily.
3. Understand that his participation is voluntary and that he is free to withdraw at any time without giving any reason, without his medical care or legal rights being affected.
4. Understand that relevant sections of his dental notes may be looked at by responsible individuals from regulatory authorities where it is relevant to his taking part in this research and give permission for these individuals to have access to his records.
5. Agree to take part in this study.
6. Participants would have the opportunity to withdraw consent at any time and to ask for their samples to be destroyed or the data excluded from research

Risk, burden, and benefits:

Those patients who consent to participate will undergo a routine dental examination to detect the dental caries extent by the aid of dental examination kit and fluorescence image evaluator device and they will be expected to collect a sample of supragingival plaque, saliva and blood.

This study is observational study without any intervention so no harm expected for these participants There may be some benefit to the participant, since they will receive full mouth examination and cleaning if required in addition to the blood test for HbAc and vitamin D level.

Confidentiality:

Confidentiality will be observed in relation to the Caldicott Principles. Only the CI and PI will have access to this information which will be coded and secured safely by password protection and encryption.

Conflict of interest:

There are no known conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* Participants may enter the trial if the following apply:
* Participants who are male or female ≥ 18 years of age.
* For the test group, they have been diagnosed with type 2 Diabetes
* For the control group, participants who are not diagnosed with type 2 Diabetes
* Particiapants having minimum one natural tooth
* They are capable of giving informed consent
* They have the ability to understand and speak English
* They are able and willing to comply with all trial requirements
* They are not participating in another dental trial
* They are not diagnosed for cognitive defect due to mental illness, depression, Alzheimer's disease, or dementia.
* No antibiotics, no steroidal and/or non-steroidal anti-inflammatory medication used during the last 3 weeks
* Participants who are not pregnant and also not breastfeeding
* Participations who are not in another dental study testing different dental products during the previous three months and during the study period
* Participants who are not currently taking Vitamin D supplements

Exclusion Criteria:

* - Participants may not enter the trial if ANY of the following apply:
* Participants who are edentulous
* Cognitive defect due to mental illness, depression, Alzheimer's disease, or dementia.
* The presence of any hard or soft tissue tumours in the oral cavity
* Patients undergoing chemo and/or radiation therapy
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Any condition, which in the opinion of the investigator, would preclude participation by the subject (such as cross-infection control risk)
* Participants who are prescribed long-term systematic antibiotics
* Participants who are pregnant and breastfeeding
* Participations who are in another dental study testing different dental products during the previous three months and during the study period
* Participants who had additional fluoride treatment in the past 6/3 months
* Participants who are prescribed to use high fluoridated toothpaste
* Participants who are currently taking Vitamin D supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For case group, Participant mainly diagnosed with diabetes mellitus type 2
  For the control group, healthy volunteer with no diabetes mellitus.
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
The extent of coronal dental caries | Initial screening
  The extent of dental caries is investigated using well-establish scoring system called "International Caries Detection and Assessment System" (ICDAS)
The extent of root dental caries | Initial screening
  The extent of root dental caries is investigated using well-establish scoring system called severity index

SECONDARY OUTCOMES:
Dental caries risk levels | Initial screening
  Dental caries risk levels is measured using Caries Management by Risk Assessment (CAMBRA)
Estimation of Cariogenic bacteria (Mutans streptococci) | Initial screening
  Estimation of Streptococcus mutans in supraginigival plaque by a real-time PCR assay
Estimation of Cariogenic bacteria (Lactobacillus ) | Initial screening
  Estimation of Lactobacillus bacteria in supraginigival plaque by a real-time PCR assay
Estimation of Cariogenic bacteria (Actinomyces) | Initial screening
  Estimation of Actinomyces bacteria in supraginigival plaque by a real-time PCR assay
Estimation of total bacterial load | Initial screening
  Estimation of total bacterial load in supraginigival plaque by a real-time PCR assay
Estimation of unstimulated saliva flow rate | Initial screening
  Estimation of unstimulated saliva flow rate by measuring saliva weight
Estimation of buffer capacity | Initial screening
  Estimation of buffer capacity using the saliva- check buffer testing mat kit
Estimation of pH | Initial screening
  Estimation of pH using the saliva- check buffer testing mat kit
Estimation Spinnbarkeit | Initial screening
  Estimation Spinnbarkeit using the NevaMeter device
Estimation of stimulated whole saliva metabolic profile. | Initial screening
  Estimation of stimulated whole saliva metabolic profile by using NMR
Estimation of saliva electrolytes | Initial screening
  Estimation of saliva electrolytes by using Inductively Coupled Plasma Optical Emission Spectroscopy (ICP-OES)
Measuring the blood HbA1c | Initial screening
  Measuring the blood HbA1c levels using point of care system
Measuring the vitamin D levels | Initial screening
  Measuring the vitamin D levels using point of care system

CONTACTS AND LOCATIONS:
Overall Officials: AShwaq Alkahtani, BSc,MSc, Principal Investigator — Queen May University of London
Locations (1):
- Royal London Dental Hospital, London, United Kingdom